CLINICAL TRIAL: NCT06776861
Title: A Prospective, Multicenter, Observational Cohort Study Assessing the Efficacy and Safety of Radiotherapy-sensitized Immunotherapy in Advanced Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, Deputy Director of the Department of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC4908
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-09

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Peripheral blood and tissue samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: PD-1 / PD-L1 monoclonal antibody — Patients with advanced breast cancer who have already received and continue to use immunotherapy, or are planned to receive immunotherapy, and have been recommended for radiotherapy after evaluation by a multidisciplinary team (MDT) in the early stage and have completed radiotherapy, are registered and followed up in this study.
  Other Names: Radiotherapy.

SUMMARY:
A prospective, multicenter, observational cohort study assessing the efficacy and safety of radiotherapy-sensitized immunotherapy in advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for inclusion in the study only if all the following criteria apply:

1. Men or women who are 18 years of age or older on the day of signing the informed consent;
2. Patients with advanced breast cancer that is inoperable or has metastasized, confirmed by histology or cytology;
3. Patients who, after MDT discussion at the metastatic breast cancer stage, are considered suitable for radiotherapy and have completed radiotherapy;
4. Patients who have previously received and continue to use immunotherapy, or are planned to receive immunotherapy, and are scheduled to receive a systemic treatment regimen including immunotherapy as chosen by the physician within 3 weeks after completing radiotherapy;
5. Patients with a traceable medical history during treatment;
6. Subjects who are able to sign an informed consent to participate in the study.

Exclusion Criteria:

1. Subjects with brain metastases or leptomeningeal metastases; if there are any suspected symptoms or signs of CNS involvement, they should be excluded by a cranial MRI scan;
2. Have not signed the informed consent form;
3. Pregnant or lactating women;
4. Other conditions deemed unsuitable for inclusion in the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced breast cancer who have already received and continue to use immunotherapy, or are planned to receive immunotherapy, and have been recommended for radiotherapy following evaluation by a multidisciplinary team (MDT) in the early stage and have completed radiotherapy, are registered and followed up in this study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2028-09-10 (Estimated); Study Completion 2028-09-10 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | 24 months
  According to RECIST 1.1 criteria：Disease Progression (PD): Referring to the smallest sum of the diameters of all measured target lesions throughout the entire experimental study, there is a relative increase of at least 20% in the sum of the diameters (if the baseline measurement is the smallest, then the baseline value is used as the reference); in addition, there must be an absolute increase of at least 5 mm in the sum of the diameters (the appearance of one or more new lesions is also considered disease progression).

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China